CLINICAL TRIAL: NCT04815226
Title: The Role of Active Administration of Peristeen Bowel Evacuation for the Management of Urinary Tract Infection in Patients With Neurogenic Bladder: a Prospective, Explorative Pilot Study
Brief Title: The Role of Active Administration of Peristeen Bowel Evacuation for the Management of Urinary Tract Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Collaborators: Coloplast A/S (Industry)
Responsible Party: Principal Investigator, Kwanjin Park, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2102-095-1198
Record Dates: First submitted 2021-03-16; First posted 2021-03-24 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Neurogenic Bladder; Neurogenic Bowel; Spina Bifida; Fecal Incontinence; Fecal Impaction; Urinary Incontinence
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Neurogenic Bowel; Spinal Dysraphism; Fecal Incontinence; Fecal Impaction; Urinary Incontinence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Using Peristeen Transanal Irrigation (Other): All participants in the trial will use Peristeen Transanal Irrigation. Eligible volunteers will be those patients who have failed conventional supportive bowel care, have neurogenic bladder, and use CIC (ClC: Clean Intermittent Catheterization) daily.
  Interventions: Device: Peristeen Transanal Irrigation

INTERVENTIONS:
Device: Peristeen Transanal Irrigation — Using Peristeen Transanal Irrigation twice per week for 12 weeks

SUMMARY:
This study investigates whether active use of transanal irrigation (Peristeen®) effectively manages urinary tract infection among patients with the diagnosis of neurogenic bladder.

DETAILED DESCRIPTION:
This study investigates whether active use of transanal irrigation (Peristeen®) effectively manages urinary tract infection among patients diagnosed with neurogenic bladder. It is a prospective exploratory pilot study, and the participants will be asked to perform transanal irrigation twice weekly for 12 weeks (three months). At each visit, including baseline, the study endpoints will be assessed by basic urinalysis, KUB imaging, Seoul Fecal Scoring, and a survey (Korean Neurogenic Bowel Score).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages, 5 to 18, and are diagnosed with neurogenic bladder.
* Use CIC (CIC: Clean Intermittent Catheterization) daily to empty the bladder.
* A recent history of fecal incontinence within the last 3 months
* More than two episodes of urinary tract infection and/ or pyuria within the last 6 months

Exclusion Criteria:

* An anatomical abnormality of the bladder neck.
* Known intractable origin of bacteriuria such as urolithiasis (kidney stone) or nonfunctional renal segment.
* Received bladder augmentation surgery
* Patient without completion of toilet training
* Either received following treatment diagnosed according to Peristeen® product safety guideline:

  1. Anorectal malformation
  2. Colorectal cancer
  3. Endoscopic polyp removal surgery in 3 months
  4. Ischemic colitis
  5. Acute inflammatory bowel disease
  6. Acute intestinal diverticulum.
  7. Radiotherapy to the colon
  8. Long-term corticosteroid usage

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in nitrite and leukocyte esterase | Baseline
  Either complete or partial reduction of nitrite and leukocyte esterase on the dip stick urinalysis
Change in nitrite and leukocyte esterase | 4 weeks
  Either complete or partial reduction of nitrite and leukocyte esterase on the
Change in nitrite and leukocyte esterase | 8 weeks
  Either complete or partial reduction of nitrite and leukocyte esterase on the
Change in nitrite and leukocyte esterase | 12 weeks
  Either complete or partial reduction of nitrite and leukocyte esterase on the

SECONDARY OUTCOMES:
Seoul Fecal Scoring | Baseline, 4 weeks, 8 weeks, 12 weeks
  Measuring the amount of feces in the abdomen using the images obtained from KUB (Kidney, Ureter, Bladder) x-ray.
Korean Neurogenic Bowel Dysfunction Score | Baseline, 4 weeks, 8 weeks, 12 weeks
  Quality of life and bowel symptom changes after using Peristeen Transanal Irrigation. 0 being having excellent quality of life and least bowel symptom changes, and 47 being the highest with extremely low QoL
Safety efficacy of Peristeen Transanal Irrigation | 4 weeks, 8 weeks, 12 weeks
  Incidence of adverse events while using Peristeen Transanal Irrigation throughout the trial using self designed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kwanjin Park, M.D. Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No